CLINICAL TRIAL: NCT02611505
Title: An Open-Label, Single-Dose, Parallel-Group Study to Assess the Effects of Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of Intranasally Administered Esketamine
Brief Title: A Study to Assess the Effects of Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of Intranasally Administered Esketamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108098; ESKETINTRD1011 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-11-19; First posted 2015-11-20 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Hepatic Impairment; Normal Hepatic Function
Keywords: Healthy; Esketamine; Hepatic Impairment; Pharmacokinetics
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants with moderate hepatic impairment will receive esketamine solution (containing 14 milligram [mg] of esketamine base per 100 microliter [mcl]) by intranasal route into each nostril using nasal spray pump at 0 hour (h) on Day 1.
  Interventions: Drug: Esketamine
- Cohort 2 (Experimental): Participants with mild hepatic impairment will receive esketamine solution (containing 14 mg of esketamine base per 100 mcl) by intranasal route into each nostril using nasal spray pump at 0h on Day 1.
  Interventions: Drug: Esketamine
- Cohort 3 (Experimental): Participants with normal hepatic function and no evidence of liver damage will receive esketamine solution (containing 14 mg of esketamine base per 100 mcl) by intranasal route into each nostril using nasal spray pump at 0h on Day 1.
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — Esketamine 28 mg will be self-administered by participants as intranasal spray at 0 hour (h) on Day 1.
  Other Names: JNJ-54135419

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety, and tolerability of intranasally administered esketamine in both participants with varying stages of hepatic impairment and healthy participants.

DETAILED DESCRIPTION:
This is a parallel group, single-center, single-dose, open-label (all people know the identity of the intervention), study to assess the pharmacokinetics and safety of a single 28 milligram (mg) dose of esketamine in both participants with varying stages of hepatic impairment and healthy participants. The participants will be assigned to 1 of 3 groups (8 participants per group) based on hepatic impairment which will be classified during Screening. Cohort 1 (participants with moderate hepatic impairment), Cohort 2 (participants with mild hepatic impairment), and Cohort 3 (participants with normal hepatic function and no evidence of liver damage). Participants will self-administer a single dose of intranasal Esketamine 28 mg. The total duration of the study from Screening through Follow-up, is approximately 34 to 38 days. Blood and urine samples for assessment of Esketamine pharmacokinetics will be collected for up to 60 hours after study drug administration. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Cohorts 1, 2 and 3 (All participants):

* Body mass index (BMI) between 18 and 34 kilogram (kg)/meter square ([m]^2) (inclusive), and body weight not less than 50 kilogram (kg)
* Creatinine clearance of greater than or equal to (> =) 60 milliliter per minute (mL/min) based on the Cockcroft-Gault equation
* Signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study

Cohorts 1 and 2 (Participants with Hepatic impairment):

* A total Child-Pugh score of 5 or 6 for participants with mild impairment and between 7 and 9 (inclusive) for participants with moderate impairment
* Participants must have stable hepatic function and consistent classification (mild or moderate hepatic impairment) between Screening and Day -1

Exclusion Criteria:

Cohorts 1, 2 and 3 (All participants):

* Participants of Asian origin
* Diagnosed with a current or previous psychotic or major depressive disorder (MDD) with psychosis, bipolar or related disorder, intellectual disability, borderline personality disorder, or antisocial personality disorder

Cohorts 1 and 2 (Participants with Hepatic impairment):

* History of hepatopulmonary syndrome, hydrothorax or hepatorenal syndrome
* Positive test for alcohol or drugs of abuse per local standard practices

Cohorts 3 (Healthy participants):

* Clinically significant medical illness
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at Screening or at admission to the study center (Day -1) as deemed appropriate by the investigator
* Positive test for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies at Screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | up to 60 hours after study drug administration
  The Cmax is the maximum plasma concentration.
Time to Reach Maximum Concentration (tmax) | up to 60 hours after study drug administration
  Time to reach the maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last (AUC [0-last]) | up to 60 hours after study drug administration
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | up to 60 hours after study drug administration
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Elimination Half-life period (t1/2) Associated with the Terminal Slope (Lambda z) | up to 60 hours after study drug administration
  Elimination half-life associated with the terminal slope (lambda[z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Area Under the Plasma Concentration-Time Curve From Time Zero to 12 Hours (AUC [0-12]) | up to 12 hours after study drug administration
  The AUC (0-12) is the area under the plasma concentration-time curve from time 0 to 12 hours post-dose.
Rate Constant (Lambda[z]) | up to 60 hours after study drug administration
  Lambda(z) is first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Cmax Metabolite to Parent Ratio (MPR Cmax) | up to 60 hours after study drug administration
  Cmax metabolite to parent ratio, and corrected for molecular weight if necessary.
AUC(last) Metabolite to Parent Ratio (MPR AUC[last]) | up to 60 hours after study drug administration
  AUC(last) metabolite to parent ratio, and corrected for molecular weight if necessary.
AUC (infinity) Metabolite to Parent Ratio (MPR AUC [infinity]) | up to 60 hours after study drug administration
  AUC (infinity) metabolite to parent ratio, and corrected for molecular weight if necessary.
Amount of Drug Excreted in Urine (Ae) | up to 60 hours after study drug administration
  Total amount excreted into the urine, calculated as the sum of all Ae(t1-t2) intervals.
Percentage of Drug dose Excreted into Urine | up to 60 hours after study drug administration
  Total amount excreted into the urine, expressed as a percentage of the administered dose, calculated as (Ae/dose)*100, and corrected for molecular weight if necessary.
Renal Clearance | up to 60 hours after study drug administration
  Renal clearance calculated as Ae/AUC (infinity).
Ae Metabolite to Parent Ratio (MPR Ae) | up to 60 hours after study drug administration
  Ae metabolite to parent ratio, and corrected for molecular weight if necessary.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to Day 11
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Knoxville, Tennessee, United States